CLINICAL TRIAL: NCT01338441
Title: Selections of Subjects With Dramatic Changes in Their Cardiac Repolarization Parameters After a Pharmacologic Stimulus Aiming to Collect Their Skin Biopsy and Blood Cells
Brief Title: Selections of Subjects With Important Changes in Their Cardiac Repolarization Parameters for the Procurement of Skin and Blood Samples
Acronym: iQTEST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ectycell SASU (Industry)
Collaborators: Pierre and Marie Curie University (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 2010-022000-41
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Cardiology: RR / QT
Keywords: Drug induced QT prolongation
MeSH Terms: interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythromycin (Experimental)
  Interventions: Drug: Erythromycin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythromycin — 4mg/Kg, IV during 20 min once
  Arms: Erythromycin
Drug: Placebo — 4mg/Kg, IV during 20 min once
  Arms: Placebo

SUMMARY:
The study main objective is to assess the changes in the ventricular repolarization (measure by the delta QTcf) after drug induced stimulation, compare to placebo, in order to identify subjects with extreme responses and collecting their skin and blood samples.

DETAILED DESCRIPTION:
An ECG is performed after a dose of sotalol on about 100 healthy subjects in order to identify about 20 extreme responders (10 high responders and 10 non responders) assessed as Delta QTcf compare to baseline. The ECG will be measured and the delta QTcf will be calculated on the 20 selected subjects in a second part of the clinical trial, cross over erythromycin/placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age
* Caucasian origin
* BMI 19 to 29 kg/m²
* Informed Consent obtained
* National Health Security Number
* Eligible for Phase I as mentioned in the national registry of healthy volunteers
* For woman: use of an effective contraceptive method

Non Inclusion Criteria:

* Asthma
* Heart Rate < 50 bpm
* Hypotension with systolic blood pressure< 100 mm Hg.
* atrioventricular block (PR interval > 200 ms)
* Known Chronic illness (hepatic, renal or cardiac impairment, etc..)
* Raynaud's phenomenon
* Drug known to prolong QT (http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm) in the last 7 days.
* All chronic treatments are forbidden exceptive : oral contraceptives, paracetamol, vitamins and comfort treatment that do not prolong the QT
* Known family or individual past history of QT prolongation or unexplained syncope
* (QTcF) > 450 ms
* QRS interval non assessable on ECG at rest or bundle-branch block, QRS > 100 ms
* Allergy to macrolide type antibiotics
* Known allergy to sotalol or lidocaine
* Positive blood pregnancy test (Inclusion visit)
* Known abnormal haemostasis
* Kaliemia< 3.5 mmol/L
* Magnesemia< 0,7 mmol/L
* Under exclusion period or participating to another clinical trial on a new medicinal product
* Creatinin clearance < 80 ml/min (Cockroft and Gault formula)
* AST-ALT >3x upper normal limit

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Prolongation of cardiac QT due to erythromycin compare to Placebo reported as Delta QTcf | 1hour and 20 minutes
  Delta QTcf is measured at H0, H0+20 minutes, and H0+1h20, on groups' erythromycin and placebo. QTcf may be adjusted based on the pharmacokinetic data to ensure time of the plasmatic pick is used.

SECONDARY OUTCOMES:
Comparison Delta QTcf eryhtromycin-sotalol | over 3 hours
  compare the effect of erythromycin and sotalol on QT prologation
Assess the effect of erythromycin Twave morphologie changes | 1hour and 20 min
  Analysis of Qwave morphologic changes

CONTACTS AND LOCATIONS:
Overall Officials: Jean Sebastien Hulot, MD, Study Director — University PMCurrie-INSERM
Locations (1):
- BIOTRIAL, Rueil-Malmaison, France

REFERENCES:
- [Derived] Stillitano F, Hansen J, Kong CW, Karakikes I, Funck-Brentano C, Geng L, Scott S, Reynier S, Wu M, Valogne Y, Desseaux C, Salem JE, Jeziorowska D, Zahr N, Li R, Iyengar R, Hajjar RJ, Hulot JS. Modeling susceptibility to drug-induced long QT with a panel of subject-specific induced pluripotent stem cells. Elife. 2017 Jan 30;6:e19406. doi: 10.7554/eLife.19406. PMID 28134617